CLINICAL TRIAL: NCT02985736
Title: An Open-Label, Study Evaluating Topicort® Topical Spray 0.25% (Desoximetasone) in Patients With Scalp Psoriasis
Brief Title: Topical Scalp Psoriasis Study Evaluating Topicort Topical Spray
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Psoriasis Treatment Center of Central New Jersey (Other)
Collaborators: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JB-02
Record Dates: First submitted 2016-10-05; First posted 2016-12-07 (Estimated); Results first posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open label (Experimental)
  Interventions: Drug: Topicort Topical Spray

INTERVENTIONS:
Drug: Topicort Topical Spray

SUMMARY:
A single center, study of 20 subjects to assess 4 weeks of therapy with Topicort® twice daily BID and 12 weeks twice daily on 2 consecutive days to patients with scalp psoriasis

DETAILED DESCRIPTION:
All patients will receive Topicort® twcie daily (BID) for 4 weeks. After week 4 patients will receive Topicort® twice weekly (on consecutive days) for 12 weeks, Patients will treat other body areas affected by plaque psoriasis with Topicort® during the study period (excludes face, groin, axilla)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults ≥ 18 years of age.
2. Diagnosis of chronic plaque-type scalp psoriasis.
3. IGA of mild or greater (scalp only) determined at screening
4. Scalp surface area of 30% or greater determined at screening
5. Able to give written informed consent prior to performance of any study related procedures.
6. Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline. FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options: hormonal contraception; intrauterine device (IUD); tubal ligation; or partner's vasectomy; Male or female condom, diaphragm with spermicide, cervical cap with spermicide, or contraceptive sponge with spermicide.
7. Subject must be in general good health (except for psoriasis) as judged by the Investigator, based on medical history, physical examination.

Exclusion Criteria:

1. <30% scalp surface area
2. Scalp Investigator global assessment (IGA) clear or almost clear at time of screening
3. Any condition, which would place the subject at unacceptable risk if he/she were to participate in the study.
4. Pregnant or breast feeding, or considering becoming pregnant during the study.
5. Use of any investigational drug within 4 weeks prior to randomization, or within 5 pharmacokinetic/pharmacodynamic half lives, if known (whichever is longer).
6. Use of oral systemic medications for the treatment of psoriasis within 4 weeks (includes, but not limited to, oral corticosteroids, methotrexate, acitretin, apremilast and cyclosporine).
7. Use of ustekinumab and/or anti-IL-17 (interleukin 17) biologic therapy within 24 weeks or other experimental or commercially available biologic immune modulator(s) within 12 weeks prior to the first IP dose.
8. Patient used other topical therapies to treat within 2 weeks of the Baseline Visit (not including permitted topical therapy for face, groin and axilla).
9. Patient received ultraviolet B, UVB phototherapy within 2 weeks of Baseline.
10. Patient received psoralen and Ultraviolet A, PUVA phototherapy within 4 weeks of Baseline.
11. Patient has a known hypersensitivity to the excipients of Topicort Spray® as stated in the label.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09; Primary Completion 2017-01-27 (Actual); Study Completion 2017-01-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from private practice dermatology
Pre-assignment Details: Of the 21 patients screened for participation, 20 subjects were enrolled to receive Open Label Topicort Topical Spray
Groups:
- Topicort Topical Spray: Topicort Topical Spray applied BID for 4 weeks followed by BID on 2 consecutive days through week 16
Period: Overall Study
Arm/Group | Topicort Topical Spray
Started | 20
Completed | 17
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Topicort Topical Spray
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 6
Age, Continuous [Mean (Full Range); unit: years] | 50 [24 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Investigator Global Assessment (Scalp Only)
Description: Scalp psoriasis severity scale (score 0-4 where 0 is no psoriasis and 4 is severe)
Time Frame: 16 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Topicort Topical Spray
Number analyzed (Participants) | 20
score on a scale | 1.59 [0 to 4]

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Topicort Topical Spray
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 9/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topicort Topical Spray (N=20)
itching (Skin and subcutaneous tissue disorders) | 3 (3)
burning (Skin and subcutaneous tissue disorders) | 5 (5)
sinusitis (Infections and infestations) | 2 (2)
worsening of psoriasis (Skin and subcutaneous tissue disorders) | 2 (2)
Infected lesion (Skin and subcutaneous tissue disorders) | 1 (1)
worsening of anxiety (Psychiatric disorders) | 1 (1)
tinea (Skin and subcutaneous tissue disorders) | 1 (1)
acne (Skin and subcutaneous tissue disorders) | 2 (2)
folliculitis (Skin and subcutaneous tissue disorders) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT02985736/Prot_SAP_000.pdf